CLINICAL TRIAL: NCT00585637
Title: Defining Optimal Doses of Vitamin D for Chemoprevention in Blacks.
Brief Title: Vitamin D for Chemoprevention
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Kimmie Ng, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 07-342; P15192 (Other: Harvard School of Public Health)
Record Dates: First submitted 2007-12-24; First posted 2008-01-03 (Estimated); Results first posted 2015-04-01 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Gastrointestinal Cancers; Prostate Cancer; Hypertension
Keywords: Vitamin D; Blacks; cancer; hypertension
MeSH Terms: conditions — Gastrointestinal Neoplasms; Prostatic Neoplasms; Hypertension; Neoplasms | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): No Vitamin D
  Interventions: Dietary Supplement: Placebo
- 2 (Active Comparator): 1000 IU of Vitamin D
  Interventions: Drug: Vitamin D
- 3 (Active Comparator): 2000 IU of Vitamin D
  Interventions: Drug: Vitamin D
- 4 (Active Comparator): 4000 IU of Vitamin D
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — Taken orally every day for three months
  Arms: 2; 3; 4
Dietary Supplement: Placebo — Placebo pill taken once daily for 3 month
  Arms: 1

SUMMARY:
This study will help us know the effects of Vitamin D pills in Blacks. The results of this study may be the first step in creating ways to prevent the risks of colon and prostate cancer. It will also help us develop ways to reduce colon cancer and prostate cancer among Blacks. This study will find out if Vitamin D pills can increase Vitamin D to healthy levels in our bodies.

DETAILED DESCRIPTION:
* Participants will be asked to answer some questions about their diet, exercise and health. In addition, participants blood pressure will be taken. These assessments will occur at baseline, 3- and 6-month appointments. At baseline only, we will measure skin tone with a tool called the Photovolt 577.
* A small blood sample will be taken to see how much Vitamin D is the body and will also look at levels of other markers of disease such as proteins, hormones, and genes.
* Participants will take a vitamin pill every day for three months and be randomly assigned to one of four different types of pills.
* Participants will be called or visited at least every two weeks. They will be asked questions to determine if they have any side effects associated with high levels of Vitamin D.
* At the beginning of the second and third months, participants will be provided with more pills. At the end of the third month, another blood sample will be taken. Three months after that, the final blood sample will be taken.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 30 and 80 years
* Comfortable communicating in English
* Currently has a primary care physician
* Willing to discontinue vitamin D or calcium supplements
* Willing to have all protocol specific tests run

Exclusion Criteria:

* Plans on taking a vacation or travel to a sunny region within 3 months of vitamin supplementation period except for a short period (i.e. 1 weekend)
* Pregnant or breast feeding or planning on becoming pregnant in the following year
* Pre-existing calcium (including hypercalcemia), parathyroid conditions (including hyperparathyroidism), sarcoidosis
* No concurrent active malignancies (other than non-melanoma skin cancer) or previous diagnosis of prostate cancer
* Cognitively impaired
* Active thyroid disease (e.g. Graves, Hashimoto's or thyroiditis)
* History of nephrolithiasis, chronic liver disease, chronic renal disease, or renal dialysis

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2007-10; Primary Completion 2010-10 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Giovannucci, MD, ScD, Principal Investigator — Harvard School of Public Health/Brigham and Women's Hospital; Gary G Bennett, PhD, Study Director — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

REFERENCES:
- [Result] Chandler PD, Scott JB, Drake BF, Ng K, Forman JP, Chan AT, Bennett GG, Hollis BW, Giovannucci EL, Emmons KM, Fuchs CS. Risk of hypercalcemia in blacks taking hydrochlorothiazide and vitamin D. Am J Med. 2014 Aug;127(8):772-8. doi: 10.1016/j.amjmed.2014.02.044. Epub 2014 Mar 20. PMID 24657333
- [Result] Ng K, Scott JB, Drake BF, Chan AT, Hollis BW, Chandler PD, Bennett GG, Giovannucci EL, Gonzalez-Suarez E, Meyerhardt JA, Emmons KM, Fuchs CS. Dose response to vitamin D supplementation in African Americans: results of a 4-arm, randomized, placebo-controlled trial. Am J Clin Nutr. 2014 Mar;99(3):587-98. doi: 10.3945/ajcn.113.067777. Epub 2013 Dec 24. PMID 24368437
- [Result] Chandler PD, Scott JB, Drake BF, Ng K, Manson JE, Rifai N, Chan AT, Bennett GG, Hollis BW, Giovannucci EL, Emmons KM, Fuchs CS. Impact of vitamin D supplementation on inflammatory markers in African Americans: results of a four-arm, randomized, placebo-controlled trial. Cancer Prev Res (Phila). 2014 Feb;7(2):218-25. doi: 10.1158/1940-6207.CAPR-13-0338-T. Epub 2013 Dec 10. PMID 24327720
- [Derived] Chandler PD, Agboola F, Ng K, Scott JB, Drake BF, Bennett GG, Chan AT, Hollis BW, Emmons KM, Fuchs CS, Giovannucci EL. Reduction of Parathyroid Hormone with Vitamin D Supplementation in Blacks: A Randomized Controlled Trial. BMC Nutr. 2015;1:26. doi: 10.1186/s40795-015-0024-8. Epub 2015 Dec 17. PMID 26858840
- [Derived] Chandler PD, Giovannucci EL, Scott JB, Bennett GG, Ng K, Chan AT, Hollis BW, Emmons KM, Fuchs CS, Drake BF. Null association between vitamin D and PSA levels among black men in a vitamin D supplementation trial. Cancer Epidemiol Biomarkers Prev. 2014 Sep;23(9):1944-7. doi: 10.1158/1055-9965.EPI-14-0522. Epub 2014 Jun 28. PMID 24974387
- [Derived] Forman JP, Scott JB, Ng K, Drake BF, Suarez EG, Hayden DL, Bennett GG, Chandler PD, Hollis BW, Emmons KM, Giovannucci EL, Fuchs CS, Chan AT. Effect of vitamin D supplementation on blood pressure in blacks. Hypertension. 2013 Apr;61(4):779-85. doi: 10.1161/HYPERTENSIONAHA.111.00659. PMID 23487599

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study recruited community-based African American (www.clinicaltrials.gov; NCT00585637). Participants were drawn from the Open Doors to Health, which is a colorectal cancer prevention study in 1554 subjects from 12 public-housing communities and community- and faith-based organizations in Boston.
Groups:
- No Vitamin D: No Vitamin D
  Placebo: Placebo pill taken once daily for 3 month
- 1000 IU of Vitamin D: 1000 IU of Vitamin D
  Vitamin D: Taken orally every day for three months
- 2000 IU of Vitamin D: 2000 IU of Vitamin D
  Vitamin D: Taken orally every day for three months
- 4000 IU of Vitamin D: 4000 IU of Vitamin D
  Vitamin D: Taken orally every day for three months
Period: Baseline
Arm/Group | No Vitamin D | 1000 IU of Vitamin D | 2000 IU of Vitamin D | 4000 IU of Vitamin D
Started | 81 | 81 | 83 | 83
Completed | 81 | 81 | 83 | 83
Not Completed | 0 | 0 | 0 | 0
Period: 3-month Time Point
Arm/Group | No Vitamin D | 1000 IU of Vitamin D | 2000 IU of Vitamin D | 4000 IU of Vitamin D
Started | 81 | 81 | 83 | 83
Completed | 71 | 67 | 76 | 78
Not Completed | 10 | 14 | 7 | 5
Period: 6-month Time Point
Arm/Group | No Vitamin D | 1000 IU of Vitamin D | 2000 IU of Vitamin D | 4000 IU of Vitamin D
Started | 81 | 81 | 83 | 83
Completed | 75 | 68 | 72 | 77
Not Completed | 6 | 13 | 11 | 6

BASELINE CHARACTERISTICS:
Population: Participants were drawn from the Open Doors to Health, which is a colorectal cancer prevention study in 1554 subjects from 12 public-housing communities and community- and faith-based organizations in Boston.
Groups:
- Total: Total of all reporting groups
Arm/Group | No Vitamin D | 1000 IU of Vitamin D | 2000 IU of Vitamin D | 4000 IU of Vitamin D | Total
Number analyzed (Participants) | 81 | 81 | 83 | 83 | 328
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 50.7 [44.2 to 58.0] | 51.1 [43.4 to 60.1] | 50.3 [43.4 to 58.2] | 51.3 [44.1 to 59.7] | 51.0 [43.6 to 59.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 59 | 55 | 54 | 222
  Male | 27 | 22 | 28 | 29 | 106
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 81 | 81 | 83 | 83 | 328
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 81 | 81 | 83 | 83 | 328

OUTCOME MEASURES:

1. Primary Outcome: Levels of Plasma 25(OH)D at Baseline, 3 Months and 6 Months.
Description: Among Blacks, identify a dose of oral vitamin D supplementation that will result in levels of plasma 25(OH)D that would be predicted to reduce colorectal cancer incidence. Community-based African Americans drawn from the Open Doors to Health, which is a colorectal cancer prevention study in 1554 subjects from 12 public-housing communities and community- and faith-based organizations in Boston.
Time Frame: Baseline, 3months, 6months
Population: Number of participants analyzed above is for baseline. At 3 months, number of participants analyzed was: 71 (no vitamin D), 67 (1000 IU Vitamin D), 76 (2000 IU Vitamin D) and 78 (4000 IU Vitamin D). At 6 months, number of participants analyzed was: 75 (no vitamin D), 68 (1000 IU Vitamin D), 72 (2000 IU Vitamin D) and 77 (4000 IU Vitamin D).
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | No Vitamin D | 1000 IU of Vitamin D | 2000 IU of Vitamin D | 4000 IU of Vitamin D
Number analyzed (Participants) | 81 | 81 | 83 | 83
ng/mL
  Baseline 25(OH)D | 15.1 [10.4 to 23.6] | 16.2 [11.0 to 22.7] | 13.9 [9.5 to 22.3] | 15.7 [11.0 to 23.3]
  25(OH)D at 3 months | 13.7 [7.2 to 18.6] | 29.7 [25.6 to 32.9] | 34.8 [28.8 to 41.0] | 45.9 [39.4 to 55.2]
  25(OH)D at 6 months | 18.1 [12.2 to 23.3] | 21.2 [16.8 to 27.8] | 27.0 [20.6 to 31.1] | 31.2 [26.5 to 35.9]

2. Secondary Outcome: Change in IL-6 From 0 to 3 Months.
Description: Examine the influence of oral vitamin D supplementation on inflammatory marker IL-6 from baseline to the 3 month follow-up.
Time Frame: From baseline to 3 months
Population: Community-based African Americans drawn from the Open Doors to Health, which is a colorectal cancer prevention study in 1554 subjects from 12 public-housing communities and community- and faith-based organizations in Boston.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | No Vitamin D | 1000 IU of Vitamin D | 2000 IU of Vitamin D | 4000 IU of Vitamin D
Number analyzed (Participants) | 71 | 67 | 76 | 78
pg/mL | -0.03 [-0.96 to 0.88] | -0.07 [-1.07 to 0.93] | 0.01 [-0.57 to 0.89] | 0.08 [-0.61 to 0.71]

3. Secondary Outcome: Change in IL-10 From 0 to 3 Months.
Description: Examine the influence of oral vitamin D supplementation on inflammatory marker IL-10 from baseline to the 3 month follow-up.
Time Frame: From baseline to 3 months
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | No Vitamin D | 1000 IU of Vitamin D | 2000 IU of Vitamin D | 4000 IU of Vitamin D
Number analyzed (Participants) | 71 | 67 | 76 | 78
pg/mL | 0 [-0.06 to 0.07] | -0.01 [-0.08 to 0.02] | -0.02 [-0.09 to 0.02] | 0.00 [-0.06 to 0.04]

4. Secondary Outcome: Change in sTNF-R2 From 0 to 3 Months.
Description: Examine the influence of oral vitamin D supplementation on inflammatory marker sTNF-R2 from baseline to the 3 month follow-up.
Time Frame: From baseline to 3 months
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | No Vitamin D | 1000 IU of Vitamin D | 2000 IU of Vitamin D | 4000 IU of Vitamin D
Number analyzed (Participants) | 71 | 67 | 76 | 78
pg/mL | -0.89 [-187.75 to 160.10] | -9.88 [-130.28 to 149.19] | 59.16 [-132.66 to 214.59] | 13.29 [-137.03 to 144.32]

5. Secondary Outcome: Change in CRP From 0 to 3 Months.
Description: Examine the influence of oral vitamin D supplementation on inflammatory marker CRP from baseline to the 3 month follow-up.
Time Frame: From baseline to 3 months
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | No Vitamin D | 1000 IU of Vitamin D | 2000 IU of Vitamin D | 4000 IU of Vitamin D
Number analyzed (Participants) | 71 | 67 | 76 | 78
mg/L | -0.05 [-1.13 to 0.98] | 0.07 [-0.58 to 0.86] | 0.02 [-0.68 to 1.21] | 0.03 [-0.68 to 0.79]

ADVERSE EVENTS:
Time Frame: Every 2 weeks, up to 6 months.
Description: Participants were assessed every 2 weeks. The table for 'Other (Non-Serious) Adverse Events' only reports on a subset of patients as calcium levels were only checked in a subset of patients. Although all patients were evaluated for adverse events, the only reported adverse event was hypercalcemia.
Arm/Group | No Vitamin D | 1000 IU of Vitamin D | 2000 IU of Vitamin D | 4000 IU of Vitamin D
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/81 | 0/83 | 0/83
Other Adverse Events (participants affected / at risk) | 0/29 | 3/28 | 1/31 | 1/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | No Vitamin D (N=29) | 1000 IU of Vitamin D (N=28) | 2000 IU of Vitamin D (N=31) | 4000 IU of Vitamin D (N=31)
hypercalcemia at 1 month (Metabolism and nutrition disorders) | 0/22 (0) | 3/23 (3) | 1/16 (1) | 0/18 (0)
hypercalcemia at 3 months (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less